CLINICAL TRIAL: NCT00053404
Title: Observational Study of HIV Infected Adults With Detectable Plasma HIV-1 RNA Levels Between 200 and 10,000 Copies/mL While Receiving Stable Antiretroviral Therapy
Brief Title: Immunologic Control of Drug Resistant HIV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Steven G. Deeks, MD, Department of Medicine, University of California - San Francisco
Other Study IDs: 1R01AI052745-01 (NIH); 1R01AI052745-01 (NIH)
Record Dates: First submitted 2003-01-28; First posted 2003-01-29 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Drug Resistance
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection

SUMMARY:
Drug resistant HIV strains often develop in patients who have taken anti-HIV drugs for an extended time. However, these drug resistant HIV strains do not always cause an increase in the level of HIV in the blood. This study will explore why some patients with drug resistant virus continue to have low viral loads.

DETAILED DESCRIPTION:
Despite the emergence of high level drug resistance in HIV-infected patients on stable antiretroviral therapy, plasma HIV RNA levels generally remain below the pretherapy viral load "set-point". The virologic and immunologic determinants of this lower steady state level of viremia have not been defined. Preliminary data indicate that: 1) drug resistant variants have reduced replicative capacity and pathogenic potential; 2) drug resistant viremia is associated with reduced T cell activation and turnover compared to wild-type viremia; and 3) patients with low level drug resistant viremia often have HIV-specific CD4 cells that are absent in patients with higher levels of viremia. This study will investigate whether the emergence of a poorly fit, drug resistant variant results in the generation of an effective HIV-specific CD4 cell response and if this response contributes to the establishment of a lower steady state level of viremia.

Participants in this study will be followed for 2 years or until antiretroviral therapy is modified or discontinued. Study visits will occur every 2 months, for a total of 14 visits. Study visits will include a patient interview and blood tests to measure the breadth and magnitude of the HIV-specific CD4 and CD8 cell responses as a function of viral load, viral replicative capacity, drug resistance phenotype, T cell turnover, and thymic function.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected for at least 6 months prior to study entry
* Documented pretherapy or off-therapy viral load of more than 10,000 copies/ml on at least 2 occasions or more than 20,000 copies/ml on at least 1 occasion
* At least a 70% reduction in plasma HIV RNA levels from pretherapy baseline
* Stable highly active antiretroviral therapy (HAART) regimen for at least 4 months prior to study entry
* HIV viral load of 200 to 10,000 copies/ml for 3 months prior to study entry
* CD4 count greater than 100 cells/mm3 and a nadir CD4 count less than 500 cells/mm3
* Virologic failure as defined by DHHS guidelines on at least one HAART regimen prior to the study entry HAART regimen
* Documented adherence to antiretroviral therapy
* Two major resistance mutations to at least two antiretroviral drug classes

Exclusion Criteria:

* Significant toxicity on current HAART regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected participants receiving antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2003-03; Primary Completion 2006-12 (Actual); Study Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven G. Deeks, MD, Study Chair — Department of Medicine, University of California - San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Result] Emu B, Sinclair E, Favre D, Moretto WJ, Hsue P, Hoh R, Martin JN, Nixon DF, McCune JM, Deeks SG. Phenotypic, functional, and kinetic parameters associated with apparent T-cell control of human immunodeficiency virus replication in individuals with and without antiretroviral treatment. J Virol. 2005 Nov;79(22):14169-78. doi: 10.1128/JVI.79.22.14169-14178.2005. PMID 16254352